CLINICAL TRIAL: NCT01862510
Title: Detection of Celiac Disease in Patients With Hypothyroidism
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Richard Zubarik, MD, University of Vermont
Other Study IDs: ZUBM12133
Record Dates: First submitted 2013-05-20; First posted 2013-05-24 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Celiac Disease; Hypothyroidism; Celiac Sprue; Malabsorption
Keywords: Celiac Disease; Hypothyroidism; Celiac Sprue; Malabsorption
MeSH Terms: conditions — Celiac Disease; Hypothyroidism; Malabsorption Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study evaluates whether hypothyroid patients requiring elevated doses of levothyroxine to maintain a euthyroid state are at increased risk of having celiac disease. It also attempts to determine if there is a threshold level of levothyroxine needed to maintain a euthyroid state in patients with hypothyroidism that should prompt serologic testing for celiac disease.

DETAILED DESCRIPTION:
This study is looking at whether hypothyroid patients who require above 125 mcg/day (or >1.5mcg/kg/day) of levothyroxine are more likely to have celiac disease than those who require smaller doses. It also looks to see if the prevalence of celiac disease in hypothyroid patients who require elevated doses of levothyroxine is high enough to warrant screening in that population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of hypothyroidism that require thyroid replacement therapy.

Exclusion Criteria:

* Surgical resection of thyroid tissue, neck irradiation, radioactive iodine therapy, prior medical treatment with lithium, methimazole, propylthiouracil, ethionamide, amiodarone, or sunitinib, prior serologic testing for celiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hypothyroidism who take thyroid replacement therapy
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
presence of celiac disease | 1 month

SECONDARY OUTCOMES:
Symptoms associated with celiac disease | 6 months
  a short questionnaire will be filled out at the time of serologic testing. If a patient hads celiac disease the form will be filled out again at 6 months after diagnosis.
medication adjustment | 6 months
  Patients diagnosed with celiac disease who initiate a gluten free diet will be assessed to determine whether adjustment of levothyroxine dosing is necessary

CONTACTS AND LOCATIONS:
Overall Officials: Richard Zubarik, MD, Principal Investigator — University of Vermont
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States

REFERENCES:
- [Background] Collins D, Wilcox R, Nathan M, Zubarik R. Celiac disease and hypothyroidism. Am J Med. 2012 Mar;125(3):278-82. doi: 10.1016/j.amjmed.2011.09.003. PMID 22340926
- [Derived] Zubarik R, Ganguly E, Nathan M, Vecchio J. Celiac disease detection in hypothyroid patients requiring elevated thyroid supplementation: A prospective cohort study. Eur J Intern Med. 2015 Dec;26(10):825-9. doi: 10.1016/j.ejim.2015.09.011. Epub 2015 Sep 28. PMID 26423749